CLINICAL TRIAL: NCT07144215
Title: ED50 of Dexmedetomidine as an Adjuvant to 0.5% Hyperbaric Bupivacaine 12.5 mg for Spinal Anesthesia in Hip and Knee Surgery: An Up-and-Down Method Approach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Raden Besthadi Sukmono, Anesthesiologist, Indonesia University
Allocation: Non-Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ED50DEXMEDETOMIDINE
Record Dates: First submitted 2025-08-20; First posted 2025-08-27 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Knee Surgery; Pelvic Surgery; Spinal Aneshtesia
MeSH Terms: interventions — Dexmedetomidine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Dexmedetomidine 3 mcg (Experimental): Patient received spinal injection of Bupivacain hyperbaric 0.5% 12.5 mg and dexmedetomidine 3 mcg.
  Interventions: Drug: Dexmedetomidine 3 mcg; Drug: Bupivacain hyperbaric 0.5% 12.5 mg
- Dexmedetomidine 4 mcg (Experimental): Patient received spinal injection of Bupivacain hyperbaric 0.5% 12.5 mg and dexmedetomidine 4 mcg.
  Interventions: Drug: Dexmedetomidine 4 mcg; Drug: Bupivacain hyperbaric 0.5% 12.5 mg
- Dexmedetomidine 5 mcg (Experimental): Patient received spinal injection of Bupivacain hyperbaric 0.5% 12.5 mg and dexmedetomidine 5 mcg.
  Interventions: Drug: Dexmedetomidine 5 mcg; Drug: Bupivacain hyperbaric 0.5% 12.5 mg
- Dexmedetomidine 6 mcg (Experimental): Patient received spinal injection of Bupivacain hyperbaric 0.5% 12.5 mg and dexmedetomidine 6 mcg.
  Interventions: Drug: Dexmedetomidine 6 mcg; Drug: Bupivacain hyperbaric 0.5% 12.5 mg

INTERVENTIONS:
Drug: Dexmedetomidine 3 mcg — Patient received spinal injection of dexmedetomidine 3 mcg.
  Arms: Dexmedetomidine 3 mcg
Drug: Dexmedetomidine 4 mcg — Patient received spinal injection of dexmedetomidine 4 mcg.
  Arms: Dexmedetomidine 4 mcg
Drug: Dexmedetomidine 5 mcg — Patient received spinal injection of dexmedetomidine 5 mcg.
  Arms: Dexmedetomidine 5 mcg
Drug: Dexmedetomidine 6 mcg — Patient received spinal injection of dexmedetomidine 6 mcg.
  Arms: Dexmedetomidine 6 mcg
Drug: Bupivacain hyperbaric 0.5% 12.5 mg — Patient received spinal injection of Bupivacain hyperbaric 0.5% 12.5 mg

SUMMARY:
Determine ED50 dexmedetomidine adjuvant that can provide spinal anesthetic sensory blockade duration of 200 minutes on knee and pelvis surgery with up-and-down method.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years old
* Pelvic or knee surgery patient with American Society of Anesthesiologists physical status I - III with epidural spinal anesthesia
* Body mass index 18-35 kg/m2
* Body height 150-180 cm
* Willing to become a research participant

Exclusion Criteria:

* Have a history of allergy to bupivacaine or dexmedetomidine
* Have sensory or motoric disabilities in the lower extremity contralateral to the surgery area
* Have a history of congestive heart failure and/or heart rhythm disorder
* Have regional anesthesia contraindication

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-05-31 (Actual); Study Completion 2025-05-31 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Effective Sensory Blockade (≥200 Minutes) | Until the end of the surgery
  Effectiveness is defined as a sensory blockade duration of at least 200 minutes from administration of spinal anesthesia with adjuvant dexmedetomidine to regression of sensory level to the T12 dermatome. Participants with blockade duration <200 minutes will be considered not effective.

SECONDARY OUTCOMES:
Hypotension Incidence | At the start of surgery until the end of surgery
  Whether the patient experienced drop in blood pressure (systolic, diastolic, and mean arterial pressure) > 20% from base value.
Bradycardia Incidence | Until the end of surgery
  Whether patient experienced drop in heart rate to <50 beat per minute.
Nausea Incidence | Until the end of surgery
  Whether patient experienced persistent nausea that cause vomiting.

CONTACTS AND LOCATIONS:
Locations (1):
- RSUPN Cipto Mangunkusumo, Jakarta Pusat, Jakarta Special Capital Region, Indonesia

IPD SHARING:
Plan to Share IPD: No